CLINICAL TRIAL: NCT01660165
Title: Mental Health and Nutritional Status During Pregnancy and Postpartum: A Prospective Study With a Nested Clinical Trial
Brief Title: Nutritional Status and Mental Health During Pregnancy and Postpartum: a Cohort Study in Rio de Janeiro, Brazil
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Gilberto Kac, Professor, Universidade Federal do Rio de Janeiro
Other Study IDs: CAAE 0139.0.314.000-09
Record Dates: First submitted 2012-05-24; First posted 2012-08-08 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Pregnancy
Keywords: Nutritional status; Mental Health; Omega-3; Pregnancy; Postpartum depression
MeSH Terms: conditions — Psychological Well-Being; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fatty acids C-reactive protein Interleukin-6
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Pregnant women

SUMMARY:
There is increasing evidence that psychosocial factors may affect health by means of biological effects and changes in behavioral health. Observational studies suggest an association between low levels of one long chain n-3 fatty acids, DHA (docosahexaenoic acid), after pregnancy and the occurrence of postpartum depression (PPD). This is an observational cohort with 4 waves of follow-up and a nested clinical trial with pregnant women residing in the city of Rio de Janeiro. The general objective is to describe the magnitude and identify factors associated to common mental disorders (CMD) during pregnancy and postpartum giving emphasis to maternal nutritional status.

Main specific objectives:

1. To evaluate the effect of CMD in the pattern of occurrence of selected maternal and child outcomes (inadequacy of gestational weight gain, postpartum weight retention, low birthweight, small for gestational weight and prematurity), considering the effect of other determinant factors, and
2. To evaluate the effectiveness of daily omega-3 doses (fish oil) in preventing PPD.

DETAILED DESCRIPTION:
The protocol predicts CMD mapping and monitoring of nutritional status throughout pregnancy and once in postpartum. Women are interviewed in four time points:

1. First trimester: 8th and 13th (baseline),
2. Second trimester: 22nd-24th gestational weeks,
3. Third trimester: 34th-36th gestational weeks,
4. Postpartum: 30-45 days

The following information will be gathered:

1. Common mental disorders (CMD): MINI International Neuropsychiatric Interview, symptoms of depression (Edinburgh scale - EPDS), anxiety (Trait Anxiety Inventory - TAI)
2. Dietary intake (food frequency questionnaire)
3. Anthropometric measure (stature and body weight) and physical activity
4. Biochemicals: fasting glucose, lipid profile (total cholesterol, HDL-c, LDL-c), serum fatty acid composition, inflammatory markers (C-reactive protein, interleukin-6), hormones (adiponectin, insulin, leptin).

All women are followed throughout pregnancy constituting the observational cohort. In the second trimester, those women identified as being in risk for PPD [past history of depression (DSM-IV) or presenting a score of depression (Edinburgh scale) >= 9 at the baseline interview] are invited to participate in the clinical trial. These women will be randomly allocated in two groups:

Intervention 1: Fish oil: [1,8 g/dia n-3 (1,08 g EPA e 0,72 g DHA)+ vit E (0,2 mg/g) Intervention 2: Placebo comparator: soybean oil + 1% fish oil + vit E (0,2 mg/g)

The supplementation occurs from the 22nd-24th week of pregnancy for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 40
* up to 13 weeks of pregnancy
* free from chronic or infectious diseases (except obesity)
* residing in the study catchment area

Exclusion Criteria:

- twin pregnancies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women attending a health care center in the city of Rio de Janeiro, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Major depressive episode | 30-45 days postpartum
  Number of women with diagnostic of major depression in the postpartum visit (30-45 days after childbirth) using Edinburgh scale and the MINI psychiatry interview.

SECONDARY OUTCOMES:
Gestational weight gain | 34-36 weeks of gestation
  Difference between last body weight measurement in pregnancy and the first assessment(8-13 weeks of gestation).
Birth weight | Postpartum
  Neonatal birth weight (grams)

OTHER OUTCOMES:
Serum fatty acids composition | 30-45 days of postpartum
  Change in n-3 (DHA, EPA) fatty acid composition (mg/dl or % of total fatty acids) throughout pregnancy and 30-45 postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Kac, Phd, Study Chair — Universidade Federal do Rio de Janeiro
Locations (1):
- Centro Municipal de Saúde Heitor Beltrão, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Vaz JDS, Farias DR, Adegboye ARA, Nardi AE, Kac G. Omega-3 supplementation from pregnancy to postpartum to prevent depressive symptoms: a randomized placebo-controlled trial. BMC Pregnancy Childbirth. 2017 Jun 9;17(1):180. doi: 10.1186/s12884-017-1365-x. PMID 28599630